CLINICAL TRIAL: NCT03393156
Title: Negative Meta-cognitions as a Causal Factor to Worry: A Randomized Controlled Trial
Brief Title: Negative Meta-cognitions as a Causal Factor to Worry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Erik Andersson, PhD, Lic. psychologist, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017/1998-31
Record Dates: First submitted 2018-01-02; First posted 2018-01-08 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Excessive Worry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-based metracognitive therapy (Experimental): The internet-based metacognitive therapy group receives a ten-week long treatment, which is based on the book "Metacognitive therapy for depression and anxiety" by Adrian Wells (2011).
  Interventions: Behavioral: Internet-based metacognitive therapy
- Wait-list (No Intervention): When the active treatment groups have finished treatment (W11), the WL group will be able to start active treatment and be assessed at post-treatment, 6 and 12 months later using the same questionnaires as the treatment group.

INTERVENTIONS:
Behavioral: Internet-based metacognitive therapy — Internet-based metacognitive therapy on a safe internet platform. Treatment is divided into ten modules, each containing homework assignments . The participants will be assigned a therapist that they can contact through a message system in the platform and expect answer within 24 hour
  Arms: Internet-based metracognitive therapy

SUMMARY:
The purpose of this study is to investigate if an internet-based metacognitive therapy reduces negative metacognitions and if reductions negative metacognitions mediates reductions in worry.

DETAILED DESCRIPTION:
The aim is primary mechanistic i.e. we want to investigate if a clear change in negative metacognitions in one group (internet-based metacognitive therapy; I-MCT) relative to another (waiting list) mediates subsequent reductions in worry.

Our hypotheses are the following:

1. I-MCT reduces both negative metacognitions (Beliefs about uncontrollability and danger of worry) and worry from baseline to week 10,
2. reductions in negative metacognitions will significantly mediate subsequent reductions in worry.

   Additionally we hypothesize that patients who score low at baseline in negative metacognitions will not show this process pattern i.e.
3. patients who score low at baseline in negative metacognitions will benefit less from treatment (moderator hypothesis)

   and consequently
4. will not show the same mediation response as stipulated in hypothesis 2 (moderated mediator hypothesis).

Trial Design: Randomized controlled trial with waitlist control. Duration: Ten weeks Primary Endpoint: Change in worry symptoms and negative metacognitions from baseline to Week 10. Long term follow-up is also investigated (baseline to 6-months after treatment completion and baseline to 12-months after treatment completion).

Efficacy Parameters: Penn State Worry Questionnaire (PSWQ) and the negative metacognitions subscale (negative beliefs about uncontrollability of thoughts and danger) of the Meta-Cognitions Questionnaire 30 items.

Safety Parameters: Adverse Events is assessed at week 10.

Description of Trial Subjects: Patients > 18 years old with a PSWQ score more than 56 points Number of Subjects: Anticipated 140

Analysis plan:

To address the hypotheses in the study growth modeling analysis using the expectation-maximization algorithm and maximum-likelihood estimation will be employed. The treatment effect on negative metacognitions and worry will examined by comparing average growth rates between treatment and control group over the assessment period. Growth modeling for longitudinal mediation will be employed to test (a) the overall mediated effect on worry using individual trajectories of change on the proposed mediator (i.e., negative metacognitions) and outcome (i.e., worry), and (b) mediated baseline by treatment moderation effect using the initial assessment of negative metacognitions as the moderator of the indirect (i.e., mediated) and direct effect of treatment. Competing mediator is depressive symptoms using the PHQ-2.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients
* ≥ 18 years
* Situated in Sweden
* Informed consent
* PSWQ score more than 56 points

Exclusion Criteria:

* Substance dependence during the last six months
* Post traumatic stress disorder, bipolar disorder or psychosis
* Symptoms better explained by axis 2 diagnosis (e.g. autism or borderline personality disorder)
* MADRS-S score above 25 points
* Psychotropic medication changes within two months prior to treatment that could affect target symptoms.
* Received metacognitive therapy for pathological worry the last 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2018-05-06 (Actual); Study Completion 2018-05-06 (Actual)

PRIMARY OUTCOMES:
Penn State Worry Questionnaire (PSWQ) | Weekly measurements week 0-10, 6 and 12 months follow-up
  Change in worry, weekly measurements, and at 6 and 12 months after treatment has ended.
Negative beliefs about uncontrollability of thoughts and danger in the Meta Cognitions Questionnaire (MCQ-30) | Weekly measurements week 0-10, 6 and 12 months follow-up
  Change in Negative beliefs about uncontrollability of thoughts and danger, weekly measurements, and at 6 and 12 months after treatment has ended.

SECONDARY OUTCOMES:
Montgomery Åsberg Depression Rating Scale (MADRS-S) | Week 0, Week 10, 6 and 12 months follow-up
  Change in depression from baseline to Week 10 and at 6 and 12 months after treatment has ended.
Euroqol, EQ-5D | Week 0, Week 10, 6 and 12 months follow-up
  Change in general health from baseline to Week 10 and at 6 and 12 months after treatment has ended
Trimbos and Institute of Medical Technology Assessment Cost Questionnaire for Psychiatry (TIC-P) [Time Frame: Week 0, Week 10, 6 and 12 months follow-up] | Week 0, Week 10, 6 and 12 months follow-up
  Change in economic costs from baseline to Week 10 and at 6 and 12 months after treatment has ended
Meta Cognitions Questionnaire (MCQ-30) | Weekly measurements, 6 and 12 months follow-up
  Change in metacognitions (all subscales as a total sum) weekly and at 6- and 12 months after treatment has ended.
Cognitive Avoidance Questionnaire (CAQ) | Week 0, Week 10, 6 and 12 months follow-up
  Change in cognitive avoidance from baseline to Week 10 and at 6- and 12 months after treatment has ended
Adverse Events | Week 10, 6 and 12 months follow-up
  Number of adverse events from baseline to Week 10 and at 6 and 12 months
Contrast avoidance questionnaire | Week 0, Week 10, 6 and 12 months follow-up
  Change in contrast avoidance from baseline to Week 10 and at 6- and 12 months after treatment has ended
Patient health questionnaire 2 items (PHQ-2) | Week 0 - Week 10 (weekly measurements), 6 and 12 months follow-up
  Change in depressive symptoms weekly measurements, and at 6 and 12 months after treatment has ended.

CONTACTS AND LOCATIONS:
Overall Officials: Erik M Andersson, PhD, Psych., Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Intitutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wahlund T, Hesser H, Perrin S, Johansson S, Huhn V, Sorhus S, Lindskog S, Serlachius E, Hedman-Lagerlof E, Ljotsson B, Andersson E. Therapist-guided online metacognitive intervention for excessive worry: a randomized controlled trial with mediation analysis. Cogn Behav Ther. 2022 Jan;51(1):21-41. doi: 10.1080/16506073.2021.1937695. Epub 2021 Jul 20. PMID 34283004